CLINICAL TRIAL: NCT03759158
Title: N-Acetyl Cysteine in the Prevention of Contrast Induced Nephropathy in Cirrhosis of Liver-NEPHRO Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-19
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Liver Cirrhoses
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC Arm (Experimental): NAC 1200 mg twice daily one day prior to the procedure and on the day of the procedure.
  Interventions: Drug: N-Acetyl Cysteine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: N-Acetyl Cysteine — NAC 1200 mg twice daily one day prior to the procedure and on the day of the procedure.
  Arms: NAC Arm
Drug: Placebo Oral Tablet — Placebo Oral Tablet twice daily.
  Arms: Placebo

SUMMARY:
Contrast induced nephropathy has an incidence of 7-11 % in patients undergoing Contrast imaging for various conditions. The risk associated with the development of CIN are still under evaluation. Even with patients having normal kidney functions there is a risk of contrast induced nephropathy hence the need for markers which could predict injury. Cirrhosis of liver predisposes patient to Kidney abnormalities as these patients lower renal reserve and can have various conditions like Hepatorenal syndrome, Sepsis, ATN. Contrast imaging is vital for ruling out conditions like Hepatocellular Carcinoma in patients of cirrhosis of liver. Presently there is no study in cirrhosis of liver which studies the Effect of N-acetyl cysteine before and after contrast imaging in the prevention Of CIN. The incidence of CNI is cirrhosis is also an avenue which requires more studies and also there is a need for formulation of a Score to predict this CIN. Hence this study is being done to assess the incidence of CNI and the role of N-Acetyl cysteine in Preventing CNI.

ELIGIBILITY:
Inclusion Criteria:

* Age-18-70 years
* Normal kidney parameters (Creatinine below <1 ,Creatinine clearance >60)
* Cirrhosis of liver
* eGFR>60ml/min

Exclusion Criteria:

* Chronic kidney disease
* H/o anaphylaxis to contrast
* Prior h/o AKI
* GFR<60 ML/MIN
* Prior H/o TACE/HVPG /Contrast ECHO in the last 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Development Of CIN (Contrast-Induced Nephropathy) (> 25% baseline creatinine) in both groups. | Day 2

SECONDARY OUTCOMES:
Mean change in serum creatinine from baseline in both groups | Day 2
Mean change in serum creatinine from baseline in both groups | Day 6
Adverse events of N-Acteyl Cysteine in both groups | Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided